CLINICAL TRIAL: NCT01895985
Title: A Single-Center, Open-Label Study Evaluating the Efficacy of Latanoprostene Bunod Ophthalmic Solution 0.024%, in Lowering Intraocular Pressure Over a 24-Hour Period in Japanese Healthy Male Volunteers
Brief Title: Efficacy of Latanoprostene Bunod in Lowering Intraocular Pressure in Japanese Healthy Male Volunteers
Acronym: KRONUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 849
Record Dates: First submitted 2013-07-03; First posted 2013-07-11 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Intraocular Pressure
MeSH Terms: interventions — BOL 303259-X

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Latanoprostene Bunod (Experimental): Participants will instill 1 drop of latanoprostene bunod 0.024% topically into each eye QD in the evening for 14 days.
  Interventions: Drug: Latanoprostene bunod

INTERVENTIONS:
Drug: Latanoprostene bunod
  Other Names: BOL-303259-X

SUMMARY:
The objective of this study is to evaluate the effect of latanoprostene bunod dosed once daily (QD) in reducing intraocular pressure (IOP) measured over a 24-hour period in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a corrected decimal visual acuity (VA) of 0.5 or better in both eyes.

Exclusion Criteria:

* Subjects with known hypersensitivity or contraindications to latanoprostene bunod, or any of the ingredients in the study drug.
* Subjects with known contraindications to NO treatment.
* Subjects who are unable to discontinue contact lens use at least 7 days prior to Visit 2 (Day 0/1/2) and during the 14 to 15-day study treatment period.
* Subjects who are unable to discontinue the use of all topical ophthalmic medications, including artificial tears, at least 7 days prior to Visit 2 (Day 0/1/2) and during the 14 to 15-day study treatment period.
* Subjects with any condition that prevents reliable applanation tonometry in either eye.
* Subjects with glaucoma in either eye.
* Subjects with any condition that prevents clear visualization of the fundus.
* Subjects who are monocular.
* Subjects with aphakia in either eye.
* Subjects with an active corneal disease in either eye.
* Subjects with severe dry eye in either eye.
* Subjects with a history/diagnosis of a clinically significant or progressive retinal disease in either eye.
* Subjects with any intraocular infection or inflammation within 3 months (90 days) prior to Visit 1 (Screening).
* Subjects with a history of ocular laser surgery within the 3 months (90 days) prior to Visit 1 (Screening).
* Subjects with a history of incisional ocular surgery or severe trauma.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
intraocular pressure (IOP) | Visit 3 (Day 14/15)
  Efficacy of latanoprostene bunod dosed QD in reducing IOP from baseline. IOP to be measured at multiple time points at visit 3.

SECONDARY OUTCOMES:
Blood levels following a single dose | 12 hours
  The systemic pharmacokinetics (PK) of latanoprostene bunod, latanoprost acid, and Butanediol Mononitrate (BDMN) following a single dose of latanoprostene bunod. blood samples to be collected pre dose, and multiple time points over a 12 hour period.
Blood levels following multiple dosing | 14 days
  The systemic PK of latanoprostene bunod, latanoprost acid and Butanediol Mononitrate (BDMN) following repeated QD dosing of latanoprostene bunod for 14 days. Blood samples to be collected prior to day 14 dose and at multiple time points following dosing over a 12 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Quintus Ngumah, OD, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Madison, New Jersey, United States

REFERENCES:
- [Result] Araie M, Sforzolini BS, Vittitow J, Weinreb RN. Evaluation of the Effect of Latanoprostene Bunod Ophthalmic Solution, 0.024% in Lowering Intraocular Pressure over 24 h in Healthy Japanese Subjects. Adv Ther. 2015 Nov;32(11):1128-39. doi: 10.1007/s12325-015-0260-y. Epub 2015 Nov 12. PMID 26563323